CLINICAL TRIAL: NCT00736593
Title: A Phase 1 Randomized, Prospective, Within-Subject, Double-Blind, Vehicle-Controlled, Dose-Escalation Study to Evaluate the Safety, Tolerability and Clinical Effect of Nexagon™ in Full-Thickness Punch Wounds
Brief Title: A Study Evaluating Nexagon™ in the Treatment of Skin Wounds.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: OcuNexus Therapeutics, Inc. (Industry)
Responsible Party: Alexis White, CoDaTherapeutics
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: NEX-SKI-001
Record Dates: First submitted 2008-08-14; First posted 2008-08-18 (Estimated); Last update posted 2009-04-27 (Estimated); Status verified 2009-04

CONDITIONS: Wound Healing
Keywords: Wound; Healing
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Nexagon™ or Nexagon™ vehicle

INTERVENTIONS:
Drug: Nexagon™ or Nexagon™ vehicle

SUMMARY:
Nexagon™ is a novel compound that promotes wound healing by temporarily disrupting cellular communication at the wound site, thereby promoting accelerated healing, reducing inflammation and pain. This randomized double-blind study will assess the safety, tolerability and clinical effect of Nexagon™ when applied to skin wounds created by punch biopsy in healthy volunteers. 43 healthy, fair-skinned males and females between ages 18-40 will be enrolled. Subjects will be reviewed again at 3 months and 9 months for follow-up safety assessments and wound appearance evaluation.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female subjects.
2. Fair skinned (Fitzpatrick Classification Level I - III).
3. Aged between 18 and 40 years inclusive.
4. Subjects who are able to comply with all study procedures, including follow-up assessment visits.
5. Subjects who are willing and able to give written informed consent to take part in the study.

Exclusion Criteria:

1. Subjects who have pigmented skin due to an increased susceptibility to hypertrophic and keloid scarring (Fitzpatrick Classification Level IV - VI).
2. Subjects who are known hypertrophic or keloid scar formers.
3. Subjects who smoke.
4. Subjects with a body mass index of greater than 30 kg/m2.
5. Subjects with bleeding disorders or taking anti-coagulants.
6. Subjects with any other skin lesion sites or a chronic or currently active skin disorder, which would adversely affect the healing of the acute wounds or which involve the areas to be examined in this study.
7. Subjects taking or who have taken prescribed drugs in the 30 days prior to Day 0, in particular, topical or systemic steroids, anti-inflammatories, anti-coagulants, anti-proliferative drugs, or antibiotics.
8. Subjects who regularly take aspirin, ginseng, gilboa, Alka Seltzer or any other over-the-counter medicine or complimentary health product that can affect the blood clotting process.
9. Subjects with a history of clinically relevant allergies.
10. Subjects with tattoos, scars or abrasions at the site to be studied.
11. Subjects with any clinically significant abnormality following review of pre-study laboratory data and physical examination.
12. Subjects showing evidence of drug abuse.
13. Subjects with any clinically significant mental illness in the opinion of the Investigator.
14. Females who are currently pregnant or breast-feeding. Females of child-bearing potential must commit to consistent and correct use of an acceptable method of birth control, as defined the protocol.
15. Subjects who have a past or present disease, which as judged by the Investigator may affect the safety of the subject or the outcome of the study.
16. Subjects who have participated in a clinical study within the 30 days prior to Day 0.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Estimated)
Dates: Start 2008-09; Primary Completion 2009-01 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Assessed by the incidence of adverse events from the time of application of the investigational product | Until the end of the study.

SECONDARY OUTCOMES:
Time to complete closure of the wounds | 35 days post-application
Rate of healing | 35 days post application
Clinical assessment by rating scales | 35 days post application
Pain | 35 days post application

CONTACTS AND LOCATIONS:
Overall Officials: Rod Ellis-Pegler, Principal Investigator — Auckland Clinical Studies
Locations (1):
- Auckland Clinical Studies, Auckland, New Zealand